CLINICAL TRIAL: NCT03905993
Title: Genetic & Environmental Determinants Of Immune Phenotype Variance: Establishing A Path Towards Personalized Medicine
Brief Title: Milieu Intérieur Collection - Genetic & Environmental Determinants Of Immune Phenotype Variance
Acronym: MI
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-070; ID-RCB : 2018-A00861-54 (Other: ANSM - Agence Nationale de Sécurité du Médicament); 10-LABX-0069 (Other Grant/Funding Number: ANR - Agence Nationale de la Recherche)
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2019-04

CONDITIONS: Individuality; Healthy Subjects
Keywords: Immune response; Immune System; genotype-to-phenotype association; genetic variability; reference-based population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. DNA extracted from whole blood
  2. Whole blood stimulations for 40 TruCulture stimulation conditions from which there are
     * Trizol stabilized cell pellets and/or extracted RNA
     * Culture supernatants in aliquots
  3. Fecal samples and extracted DNA
  4. Nasal swab samples, extracted DNA and liquid supernatant
  5. Plasma from whole blood
  6. Frozen PBMCs
  7. Fibroblast cell lines (322 donors) and derived iPSCs (4 donors)
  8. EBV cell lines (203 donors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: unique group.: At V0: 1238 subjects were screened At V1: 1012 subjects (12 later withdrew) gave the following samples: blood, nasal swab,stool. 323 subjects among 1000 gave one additional sample (Skin Biopsy) At V2: 504 subjects came at V2 to perform blood, nasal swab and stool samples

SUMMARY:
The purpose of this study is to assess the determinants of immunologic variance within the general healthy population.

DETAILED DESCRIPTION:
Susceptibility to infections, disease severity, and response to medical therapies and vaccines are highly variable from one individual to another. While the question of variance in human populations continues to be a focal point of scientific research, medical practices and public health policies typically take a 'one size fits all' model to disease management and drug development.

Individual heterogeneity in the immune response can have an enormous impact on the likelihood to respond to therapy or the development of side effects secondary to vaccine administration. Because of the complexity of immune responses in the individual and within the population, it has not been possible thus far to define the parameters (genetic or environmental) that constitute a healthy immune system and its natural occurring variability.

Efforts to restore the 'personal' in medical care are the current challenge, and the driving vision of the project, to which the current study belongs.

In order to realize the promise of personalized medicine, an in-depth understanding of the determinants of heterogeneity in host response to stress is required. The Milieu Interieur cohort was established to address these questions through a population systems immunology approach.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects considered as healthy by the investigator based on medical history, clinical examination, laboratory results and ECG (blood sampling for laboratory assessments and ECG were performed at V0 and only after signed informed consent).
2. Subjects who, according to the investigator, complied with the requirements of the protocol and were available for all scheduled visits at the investigational site.
3. Healthy male or female aged between 20 and 69 (included) years
4. Metropolitan French origin for 3 generations
5. 18.5 ≤BMI ≤ 32 kg/m²
6. Ability to give their informed consent in writing
7. Understanding of spoken and written French
8. Affiliated to the French social security or assimilated regimens

Exclusion Criteria:

1. Participation in another clinical study in the previous 3 months in which the subject had been exposed to an investigational product (pharmaceutical product or placebo or medical device) or concurrent participation in another clinical study during the study period
2. Relatedness to previously recruited individuals in the study cohort
3. Travel in (sub-)tropical countries within the previous 3 months
4. For women: pregnant or breastfeeding or intending to become pregnant or peri-menopausal*

   * Peri-menopausal women as defined by menstrual irregularity: either a change in the menstrual cycle length of more than seven days (early perimenopause) or two or more missed periods with an interval of 60 days or more between periods (late perimenopause) (Stages of Reproductive Aging Workshop, STRAW)
5. Any physical exercise within the previous 8 hours before study visits.
6. Subjects following a special diet for medical reasons as prescribed by a GP or dietician (e.g. calorie restricted or weight-loss diet for significant overweight, cholesterol lowering diet or subjects suffering from any clinically diagnosed food allergy or intolerance)
7. Alcohol abuse (more than 50 g of pure ethanol per day: for example, more than 4 x 150 mL glasses of wine, more than 4 x 250 mL glasses of beer, more than 4 x 40 mL glasses of high alcohol content drinks)
8. Illicit drug use or substance abuse within 3 months prior to inclusion
9. Presence of evidence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to participate in the study satisfactorily.
10. Severe/chronic/recurrent pathological conditions, among them:

    10.1. Past or present diagnosed cancer, lymphoma, leukemia to the exception of:
    * Persons with a history of cancer who are disease-free without treatment for 5 years or more
    * Women who are disease free for 3 years or more after treatment for breast cancer and receiving long-term prophylactic tamoxifen
    * Cutaneous or cervical basal cell carcinoma 10.2. Personal history of organ transplant 10.3. Congenital or acquired immune deficiency (any confirmed or suspected immunosuppressive or immunodeficient condition, including history of HIV infection) 10.4. Personal history of auto-immune diseases requiring or having previously required treatment (e.g. Rheumatoid Arthritis, Systemic Lupus Erythematosus, Sarcoidosis, Ankylosing Spondylitis, Autoimmune Hemolytic Anemia, Autoimmune Thrombocytopenic Purpura, Crohn's Disease, Psoriasis, Scleroderma, Wegener's Granulomatosis,Type I Diabetes, Thyroiditis,….) 10.5. Splenectomy 10.6. Acute or chronic, clinically significant, as determined by the investigator, pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests 10.7. History of clinically significant, as determined by the investigator, neurological disorder or seizures 10.8. Infectious diseases:
    * Chronic infection (e.g. HIV, HBV, HCV…) or current acute infection or past acute infection based on investigator's judgment within the previous 3 months,
    * Presence of a rectal temperature ≥38.4°C, or axillary temperature ≥37.5°C, or intra-auricular temperature ≥38.4 °C, or buccal temperature ≥38°C on the scheduled date of inclusion,
    * Subject receiving (currently or in the last 3 months) antibiotics, intestinal, nasal or respiratory antiseptics.

    10.9. Severe High Blood Pressure defined as systolic BP≥160 mmHg and/or diastolic BP≥100 mmHg (AHA stage 2 HBP). Treated and controlled HBP is allowed.

    10.10. Type II diabetes mellitus requiring treatment with any medication. Diabetes mellitus treated by exercise and diet control only is permitted.

    10.11. Chronic renal impairment as defined by Renal Insufficiency: GFR<60 mL/min/1.73 m² (National Kidney Foundation (2002).

    10.12. Chronic bone disease as treated by biphophonates. 10.13. Treated depression or any evidence of overt depressive episode during medical examination and interview.

    10.14. Any significant disorder of coagulation or treatment with warfarin derivatives or heparin or antiplatelet medications within 2 months preceding inclusion.

    10.15. Dermatologic conditions: any current dermatological disorder that is severe enough to prevent the skin biopsy (e.g. eczema, psoriasis, acute or chronic dermatitis).

    10.16. Severe acute/chronic allergy
    * Severe Asthma defined as asthma requiring a combination of two or more controller therapies (e.g. medium or high dose inhaled glucocorticosteroid and long-acting inhaled beta-2 agonist) or requiring oral glucocorticosteroids (GINA).
    * Severe food allergy, as defined by history of giant urticaria, Quincke edema or anaphylactic shock,
    * Severe insect bite allergy with history of giant urticaria, Quincke edema or anaphylactic shock,
    * Atopic dermatitis treated with medication.
11. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within the 6 months prior to the inclusion. For corticosteroids, this will mean a dose equivalent to 20 mg/day of prednisone or equivalent for > 2 weeks (inhaled and topical steroids allowed)
12. Chronic administration of NSAIDs, including aspirin: prolonged intake (> 2 weeks) within 6 months before study or any intake within the 7 days preceding skin biopsy [exception for low dose aspirin: maximum 250mg/daily, see 8.1]
13. Receipt of any vaccination 3 months before the inclusion or planning to receive any vaccination during the study
14. Receipt of blood products or immunoglobulins within 3 months prior the inclusion or planning to receive blood products or immunoglobulins during the study
15. Hemoglobin measurement less than 10.0 g/dL for women and less than 11.5 g/dL for men
16. Platelet count less than 120.000/mm3
17. ALAT and/or ASAT > 3 times the upper limit of the norm (ULN)
18. Allergy to lidocaine

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults subjects, aged from 20 to 69 years old, and whose ancestry for three generations was of Metropolitan French origin
Sampling Method: Non-Probability Sample
Enrollment: 956 (Actual)
Dates: Start 2012-09-17 (Actual); Primary Completion 2013-08-08 (Actual); Study Completion 2013-08-08 (Actual)

PRIMARY OUTCOMES:
Identify genetic associations with immune response variability | 2024
  Genome wide associations studies that combine whole genome genotyping data sets with immune response phenotypes to identify genetic regulators of immune function. These studies will be later completed with data from whole genome sequencing for more detailed genetic analysis.

SECONDARY OUTCOMES:
Identify environmental associations with immune response variability | 2026
  Association of whole metagenomic data sets generated from fecal samples that reflect environmental exposures with immune response phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Lluis Quintana-Murci, PhD, Principal Investigator — Institut Pasteur

IPD SHARING:
Plan to Share IPD: Yes
Milieu Intérieur clinical data (CRF) have already been collected, and upon publication in peer reviewed journals certain biological data sets will be deposited in secure data warehouses to allow access for scientific research use only. All MI data sets are completely pseudo-anonymized (donors' identity is replaced with a unique MI number).
  Of the 1,000 subjects enrolled in the MI study, 956 have consented for their data to used outside the consortium for scientific research use only. This usage in approved scientific collaborations is reviewed by the Milieu Interieur data and sample access committee and also covers the deposit of pseudo-anonymized data sets in centrally controlled data repositories.
  All IPD that underlie results in peer reviewed publications may be shared for scientific collaborations following a request and review by the Milieu Interieur data and sample access committee.
Supporting Information: CSR, Analytic Code
Time Frame: Until April 2028
Access Criteria: All IPD that underlie results in peer reviewed publications may be shared for scientific collaborations following a request and review by the Milieu Interieur data and sample access committee.
URL: http://www.milieuinterieur.fr

REFERENCES:
- [Background] Patin E, Hasan M, Bergstedt J, Rouilly V, Libri V, Urrutia A, Alanio C, Scepanovic P, Hammer C, Jonsson F, Beitz B, Quach H, Lim YW, Hunkapiller J, Zepeda M, Green C, Piasecka B, Leloup C, Rogge L, Huetz F, Peguillet I, Lantz O, Fontes M, Di Santo JP, Thomas S, Fellay J, Duffy D, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. Natural variation in the parameters of innate immune cells is preferentially driven by genetic factors. Nat Immunol. 2018 Mar;19(3):302-314. doi: 10.1038/s41590-018-0049-7. Epub 2018 Feb 23. PMID 29476184
- [Background] Piasecka B, Duffy D, Urrutia A, Quach H, Patin E, Posseme C, Bergstedt J, Charbit B, Rouilly V, MacPherson CR, Hasan M, Albaud B, Gentien D, Fellay J, Albert ML, Quintana-Murci L; Milieu Interieur Consortium. Distinctive roles of age, sex, and genetics in shaping transcriptional variation of human immune responses to microbial challenges. Proc Natl Acad Sci U S A. 2018 Jan 16;115(3):E488-E497. doi: 10.1073/pnas.1714765115. Epub 2017 Dec 27. PMID 29282317
- [Background] Thomas S, Rouilly V, Patin E, Alanio C, Dubois A, Delval C, Marquier LG, Fauchoux N, Sayegrih S, Vray M, Duffy D, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. The Milieu Interieur study - an integrative approach for study of human immunological variance. Clin Immunol. 2015 Apr;157(2):277-93. doi: 10.1016/j.clim.2014.12.004. Epub 2015 Jan 3. PMID 25562703
- [Background] Clave E, Araujo IL, Alanio C, Patin E, Bergstedt J, Urrutia A, Lopez-Lastra S, Li Y, Charbit B, MacPherson CR, Hasan M, Melo-Lima BL, Douay C, Saut N, Germain M, Tregouet DA, Morange PE, Fontes M, Duffy D, Di Santo JP, Quintana-Murci L, Albert ML, Toubert A; Milieu Interieur Consortium. Human thymopoiesis is influenced by a common genetic variant within the TCRA-TCRD locus. Sci Transl Med. 2018 Sep 5;10(457):eaao2966. doi: 10.1126/scitranslmed.aao2966. PMID 30185651
- See also: Related Info — http://www.milieuinterieur.fr